CLINICAL TRIAL: NCT01014715
Title: Preoperative Accelerated Partial Breast Irradiation (APBI) for Women With Stage I and Select IIA Breast Cancer
Acronym: GCC 0919
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Prinicipal Investigator, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HP-00042098; GCC 0919
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): Phase II-Preoperative Radiation followed by Lumpectomy
  Interventions: Other: Phase II - Preoperative Radiation followed by Lumpectomy.

INTERVENTIONS:
Other: Phase II - Preoperative Radiation followed by Lumpectomy. — Sequential investigative question. All procedures are standard of care

SUMMARY:
The purpose of this study is to examine the feasibility to deliver PBI before the lumpectomy is performed. By administering the PBI before the lumpectomy, a smaller volume of breast tissue may be exposed to radiation. The PBI method used in this study is 3D (three dimensional) conformal external beam irradiation. 3D-conformal external beam irradiation uses an x-ray beam to deliver the radiation dose. Approximately 3 weeks after completion of the PBI, the cancer will be surgically removed.

This study will learn about the good and bad effects of 3D-conformal external beam irradiation PBI when given before the cancer has been removed by lumpectomy. The study will also learn about the feelings women have about how their breast looks after PBI and surgery.

DETAILED DESCRIPTION:
This study will evaluate the feasibility, cosmetic results, complication rates, and local control rate of 3D-CRT confined to the region of the lumpectomy cavity for patients with Stage I and IIa (less than or equal to 3 cm) carcinoma of the breast (non-lobular histology) treated with APBI using 3D-CRT before lumpectomy. For selected patients with Stage I and II breast carcinoma, 3D-CRT delivered to the primary tumor preoperatively is technically reproducible with acceptable complication rates. Cosmetic results after partial breast irradiation before lumpectomy will be comparable to that obtained after whole breast external beam radiation therapy. The local tumor control rate in the breast after partial breast irradiation therapy followed by lumpectomy will be comparable to that of conventional external beam radiation therapy, with less inconvenience and potentially less cost to the patient, given the selection criteria which minimize the risk of clinically significant multicentric or extensive residual carcinoma following lumpectomy.

ELIGIBILITY:
Inclusion Criteria:

Women who satisfy all of the following conditions are the only patients who will be eligible for this study:

1. Patient must have invasive ductal, medullary, papillary, colloid (mucinous), or tubular histologies.
2. AJCC Stage I or IIA (T1N0 or T2N0) histologically confirmed invasive carcinoma of the breast with a primary lesion (less than/equal to 3 cm)by MRI or ultrasound
3. Clinically negative axillary lymph nodes. Standard routine imaging assessment of the axilla is performed by either ultrasound or MRI. If lymph nodes are suspicious, a biopsy is required. An involved axilla is purposely excluded.
4. Unifocal breast cancer (single focus which can be encompassed by one lumpectomy).
5. Patients must have an estrogen receptor (ER), progesterone receptor (PR), and human epidermal growth receptor 2 (H2N) analyses performed on the primary tumor prior to enrollment.
6. Based on pre-treatment planning CT scan, the ratio of the PTV to the reference breast volume should not exceed 25%.
7. Patients must be greater than/equal to 18 years of age.
8. Pretreatment evaluations required for eligibility include: bilateral mammogram, histologic confirmation of malignancy, and physical exam.
9. Signed study-specific informed consent form prior to study entry.
10. Women of childbearing potential must use an effective contraceptive method such as condom/diaphragm and spermicidal foam, intrauterine device (IUD), or prescription birth control pills.

Exclusion Criteria:

Men are not eligible for this study. Women with one or more of the following conditions also are ineligible for this study:

1. Evidence of suspicious microcalcifications which are separate from the known lesion unless pathologically confirmed to be benign.
2. Patient with distant metastases.
3. Patients with invasive lobular or extensive in-situ lobular carcinoma or pure ductal carcinoma in-situ or non-epithelial breast malignancies such as sarcoma or lymphoma.
4. Patients with proven multicentric carcinoma (tumors in different quadrants of the breast or tumor separated by at least 4 cm) or with other clinically or radiographically suspicious areas in the ipsilateral breast unless confirmed to be negative for malignancy by biopsy.
5. Patient whose tumor is not visible on radiation treatment planning CT scan
6. Palpable or radiographically suspicious ipsilateral axillary, supraclavicular, infraclavicular or internal mammary nodes, unless there is histologic confirmation that these nodes are negative for tumor.
7. Prior hormonal or non-hormonal therapy or radiation therapy for the current breast cancer.
8. Patients with Paget's disease of the nipple.
9. Patients with skin involvement, regardless of tumor size.
10. Patients with a breast technically unsatisfactory for radiation therapy.
11. Patients with collagenous diseases, specifically systemic lupus erythematosis, scleroderma, or dermatomyositis.
12. Patients with co-existing medical conditions with life expectancy less than 2 years.
13. Patients with psychiatric or addictive disorders that would preclude obtaining informed consent.
14. Patients who are pregnant or lactating due to potential exposure of the fetus to RT and unknown effects of RT to lactating females.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2018-11-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is determination of the reproducibility of delivering preoperative APBI in Stage I and Stage IIA breast cancers. | 5 years
  This will be done by using 3D-CRT by evaluating the prescription isodose curves, dose inhomogeneity, and coverage of the volume as defined by CT treatment planning to delineate the target volume.

SECONDARY OUTCOMES:
Evaluation of pathologic response, cosmetic results, of lumpectomy wound healing and the overall complication rate, ipsilateral breast recurrence rate | 5 years
  These endpoints will be accomplished by utilizing the pathology report; the cosmesis will be judged by the patient, radiation oncologist and/or surgeon, at stated follow-up intervals; and the breast recurrence rate will be evaluated by disease status at routine patient follow-up appointments, including yearly mammography.

CONTACTS AND LOCATIONS:
Overall Officials: Wendla Citron, MD, Principal Investigator — UMMC MSGCC Department of Radiation Oncology
Locations (3):
- United States (3):
  - Ummc Msgcc, Baltimore, Maryland
  - Central Maryland Oncology Center, Columbia, Maryland
  - Baltimore Washington Medical Center, Glen Burnie, Maryland